CLINICAL TRIAL: NCT04175249
Title: Effects of a Pizza Meal Challenge on the Immunometabolism of Monocytes and T Cells
Brief Title: Pizza Meal Challenge and Immunometabolism (PIMETA)
Acronym: PIMETA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Anja Maehler, Principal Investigator, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PIMETA
Record Dates: First submitted 2019-11-21; First posted 2019-11-22 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: Salt challenge; Immune cell metabolism; Oxygen consumption rate; Extracellular acidification rate; Cytokine production

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pizza meal challenge (Experimental): Vegetarian pizza containing 10 grams of salt
  Interventions: Other: Pizza meal challenge

INTERVENTIONS:
Other: Pizza meal challenge — Vegetarian pizza containing 10 grams of salt

SUMMARY:
High salt intake is a major risk factor for cardiovascular events, including stroke, heart disease and kidney failure. Pizza is a popular salty food. In this exploratory pilot study, the effects of a pizza meal challenge on immunometabolism in healthy subjects will be tested.

ELIGIBILITY:
Inclusion Criteria:

- Healthy men and women

Exclusion Criteria:

* Severe, manifest illnesses in need of treatment
* Pathological lab results
* Inability to understand significance and scope of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption rate of immune cells | 3 hours after the pizza compared to baseline
  OCR (pmol oxygen/min/1000 cells) measured by Seahorse

SECONDARY OUTCOMES:
Oxygen consumption rate of immune cells | 3 and 8 hours after the pizza adjusted for plasma sodium concentration compared to baseline
  OCR (pmol oxygen/min/1000 cells) measured by Seahorse
Plasma sodium | 3 and 8 hours after the pizza compared to baseline
  Plasma sodium concentration (mmol/l)
Mitochondrial membrane potential of immune cells | 3 and 8 hours after the pizza compared to baseline
  Mitochondrial membrane potential (Mean Fluorescence Intensity of TMRE) measured by flow cytometry
Extracellular acidification rate of immune cells | 3 and 8 hours after the pizza compared to baseline
  ECAR (mpH/min/1000 cells) measured by Seahorse
Interleukin 17 release after monocyte and T cell co-culture | Cell isolation at baseline and 3 hours after the pizza followed by 72 hours of co-culture
  IL-17 concentration (pg/ml) measured by ELISA
Interferon-gamma release after monocyte and T cell co-culture | Cell isolation at baseline and 3 hours after the pizza followed by 72 hours of co-culture
  INF-g concentration (pg/ml) measured by ELISA
Adenosine triphophate production of immune cells | 3 and 8 hours after the pizza compared to baseline
  Percent change of luminescence (%) measured by Luminescence Assay

CONTACTS AND LOCATIONS:
Overall Officials: Dominik N. Müller, PhD, Principal Investigator — Charite University, Berlin, Germany; Anja Mähler, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Experimental & Clinical Research Center, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of reported articles (text, tables, figures, supplemental data) will be shared after deidentification.
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Result] Geisberger S, Bartolomaeus H, Neubert P, Willebrand R, Zasada C, Bartolomaeus T, McParland V, Swinnen D, Geuzens A, Maifeld A, Krampert L, Vogl M, Mahler A, Wilck N, Marko L, Tilic E, Forslund SK, Binger KJ, Stegbauer J, Dechend R, Kleinewietfeld M, Jantsch J, Kempa S, Muller DN. Salt Transiently Inhibits Mitochondrial Energetics in Mononuclear Phagocytes. Circulation. 2021 Jul 13;144(2):144-158. doi: 10.1161/CIRCULATIONAHA.120.052788. Epub 2021 Apr 28. PMID 33906377